CLINICAL TRIAL: NCT05702047
Title: Comparing Nose & Mouth Breathing During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph Watso, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00003661
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nose-only breathing (Active Comparator): Participants will be instructed to breathe only through their nose (mouth closed) during rest and submaximal exercise.
  Interventions: Behavioral: Nose-only breathing
- Mouth-only breathing (Active Comparator): Participants will be instructed to breathe only through their mouth (nose clips prevent nose breathing) during rest and submaximal exercise.
  Interventions: Behavioral: Mouth-only breathing

INTERVENTIONS:
Behavioral: Nose-only breathing — Participants will breathe only through their nose (mouth closed) during rest and submaximal exercise.
  Arms: Nose-only breathing
Behavioral: Mouth-only breathing — Participants will breathe only through their mouth (nose clips prevent nose breathing) during rest and submaximal exercise.
  Arms: Mouth-only breathing

SUMMARY:
The purpose of this study is to compare physiological responses in cardiovascular variables between nose and mouth breathing at rest and during exercise.

DETAILED DESCRIPTION:
Breathing patterns can affect the cardiovascular system. Little is known about how nose versus mouth breathing affects cardiovascular variables (blood pressure, heart rate, etc.) at rest and during exercise. It has been suggested that breathing through the nose can cause calmness and lower blood pressure. However, research is needed to examine the extent to which breathing through the nose affects cardiovascular variables at rest and during exercise. Therefore, we will compare cardiovascular variables between nose-only and mouth-only breathing. The rate of breathing will be fixed (using an audible metronome) for both breathing conditions (nose-only vs mouth-only) based on an individual's free breathing (i.e., no breathing cues) breathing rate.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index: ≤30 kg/m2
* Resting Blood pressure: ≤140/90 mmHg

Exclusion Criteria:

* Overt cardiovascular (e.g., diagnosed hypertension), respiratory, neurological, renal, liver, and/or metabolic health condition
* Current or recent (regular use within the past 6 months) use of tobacco or nicotine products (e.g., cigarettes)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Watso, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate data and/or material transfer agreement approvals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completion of the trial, indefinitely
Access Criteria: A formal plan identifying the intended use of the data and proper completion of appropriate data and/or material transfer agreement approvals with the study PI and their institution.

REFERENCES:
- See also: Related Info — https://caplaboratory.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mouth Breathing Then Nose Breathing: 1. Participants will be instructed to breathe only through their mouth (nose clips on) during rest and submaximal exercise. 2. Participants will be instructed to breathe only through their nose (mouth closed) during rest and submaximal exercise.
- Nose Breathing Then Mouth Breathing: 1. Participants will be instructed to breathe only through their nose (mouth closed) during rest and submaximal exercise. 2. Participants will be instructed to breathe only through their mouth (nose clips on) during rest and submaximal exercise.
Period: Overall Study
Arm/Group | Mouth Breathing Then Nose Breathing | Nose Breathing Then Mouth Breathing
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: These numbers are for all participants
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Body mass index [Mean (Standard Deviation); unit: kilograms per meters squared] | 23 (2)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure During Exercise Between Study Arms
Description: Systolic blood pressure will be measured in the laboratory during submaximal exercise with nose-only breathing and mouth-only breathing.
Time Frame: Up to one day
Population: 17 participants completed both arms with this variable measured
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nose-only Breathing | Mouth-only Breathing
Number analyzed (Participants) | 17 | 17
mmHg | 142 (14) | 146 (12)

2. Primary Outcome: Heart Rate During Exercise Between Study Arms
Description: Heart rate will be measured in the laboratory during submaximal exercise with nose-only breathing and mouth-only breathing.
Time Frame: Up to one day
Population: 18 participants completed both arms with this variable measured
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Nose-only Breathing | Mouth-only Breathing
Number analyzed (Participants) | 18 | 18
beats per minute | 130 (20) | 133 (22)

3. Secondary Outcome: Rating of Perceived Exertion During Exercise Between Study Arms
Description: Participants will report their rating of perceived exertion (numerical scores of 6-20, with 20 being the greatest exertion) based on a validated scale during submaximal exercise with nose-only breathing and mouth-only breathing.
Time Frame: Up to one day
Population: 18 participants completed both arms with this variable measured
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nose-only Breathing | Mouth-only Breathing
Number analyzed (Participants) | 18 | 18
units on a scale | 13 (3) | 12 (2)

4. Secondary Outcome: Rating of Perceived Breathlessness During Exercise Between Study Arms
Description: Participants will report their rating of perceived breathlessness (numerical scores of 0-10, with 10 being the greatest breathlessness) based on a validated scale during submaximal exercise with nose-only breathing and mouth-only breathing.
Time Frame: Up to one day
Population: 18 participants completed both arms with this variable measured
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Nose-only Breathing | Mouth-only Breathing
Number analyzed (Participants) | 18 | 18
units on a scale | 2 [1.25 to 2.75] | 3 [1.85 to 4.15]

ADVERSE EVENTS:
Time Frame: Up to one day
Description: Participants completed both arms
Arm/Group | Nose-only Breathing | Mouth-only Breathing
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT05702047/Prot_000.pdf